CLINICAL TRIAL: NCT07306793
Title: The Effect of Oral Motor Intervention and Chronobiological Approach to Feeding Models Applied to Preterm Infants on Infants' Readiness to Feed, Transition to Total Oral Feeding, and Body Weight
Brief Title: The Effect of PIOMI and Chronobiological Nutrition on Readiness for Feeding, Full Transition to Oral Feeding and Body Weight
Acronym: PIOMI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Esra Bozkurt, MSc, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Interventional trial
Record Dates: First submitted 2025-12-13; First posted 2025-12-29 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Neonatal İntensive Care; Nutrition With A Chronobiological Approach; Readiness For Feding; Body Weight; Breast Milk; Nutrition; Premature Birth
Keywords: Neonatal İntensive Care; Nutrition With A Chronobiological Approach; Readiness For Feding; Body Weight; Transitioning To Total Oral Feeding; Premature Infant Oral Motor Intervention (PIOMI); Prematüre
MeSH Terms: conditions — Body Weight; Premature Birth | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled experimental study. There are three groups: the PIOMI study group, the chronobiological feeding model study group, and a control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PIOMI study group (Experimental): Premature infant group undergoing Oral Motor Intervention.
  Interventions: Other: PIOMI study group
- Nutrition Study Group with a Chronobiological Approach (Experimental): Group of infants fed using chronobiological approaches
  Interventions: Other: Nutrition Study Group with a Chronobiological Approach
- No Intervention (Other): Control group.
  Interventions: Other: Control group

INTERVENTIONS:
Other: PIOMI study group — Infants will be weighed at 8:30 AM wearing only a clean diaper, and the scale will be disinfected before and after each use. Preterm infants in this group will receive PIOMI treatment at their bedside for 5 minutes, once a day, 15 minutes before feeding times at 9:00 AM or 12:00 PM, for 14 days. Before starting the PIOMI treatment, the researcher will remove any jewelry and wash their hands hygienically. Following the PIOMI treatments, infants will be fed using the feeding method applied in the clinic, and this will be recorded. Infants will be monitored throughout their stay in the NICU.
  Arms: PIOMI study group
Other: Nutrition Study Group with a Chronobiological Approach — Newborns will be weighed at 8:30 a.m. wearing only a clean diaper, and the scale will be disinfected before and after each use. The researcher will provide training to the baby's mother on breast milk expression and storage. Breast milk storage bags and adhesive labels labeled "NIGHT MILK" and "DAY MILK" will be provided by the researcher. Mothers will be asked to express milk between 06:00 and 17:59, place it in a breast milk storage bag, attach the "DAY MILK" label, and write their name, surname, date, and time on it. For milk expressed between 18:00 and 05:59, they will place it in a breast milk storage bag, attach the "NIGHT MILK" label, and write their name, surname, date, and time on it, and bring their milk to the unit in this manner. Newborns in this group will be fed using breast milk that is chronobiologically matched.
  Arms: Nutrition Study Group with a Chronobiological Approach
Other: Control group — Newborns will be weighed at 8:30 AM wearing only a clean diaper, and the scale will be disinfected before and after each use. No procedures will be performed on these infants outside of the clinical routine. Infants will be fed using the same feeding method as in the clinic. Infants will be monitored throughout their stay in the NICU.
  Arms: No Intervention

SUMMARY:
This is a randomized controlled experimental study evaluating the effects of oral motor intervention and chronobiological approach to feeding model applied to preterm infants on feeding readiness, transition to total oral feeding and body weight.

DETAILED DESCRIPTION:
Premature birth is defined as birth occurring before the 37th week of gestation, and approximately 15 million babies are born this way worldwide each year. Premature babies experience feeding difficulties because their oral feeding skills, sucking-swallowing-breathing coordination, and oral structures are not fully developed. Their oral motor systems typically mature between 32-34 weeks of gestation. The development of the oral motor system is crucial for adequate nutrition, growth, and weight gain. Several methods are used to improve the oral motor development of premature babies. Oral motor interventions involve physical stimuli applied to intraoral structures such as the lips, tongue, cheeks, gums, and palate. These methods aim to increase the functional strength of oral muscles and target neuro-behavioral synergy.

Oral motor interventions applied in NICUs have been shown to accelerate the transition to oral feeding, increase weight gain, and shorten hospital stays in premature infants. Premature Infant Oral Motor Intervention (PIOMI) is one of the interventions applied in NICUs. Studies have shown that PIOMI is more effective than other interventions in this field. Furthermore, no negative side effects of PIOMI have been reported.

Breast milk is an ideal source of nutrition for the growth and development of preterm infants. It provides essential nutrients for the baby's growth and development, as well as containing biological cues that help regulate circadian rhythms. For the fetus, which has become accustomed to the mother's circadian rhythms during intrauterine life, it supports this transition process by providing similar cues after birth. The composition of breast milk can vary depending on gestational age, lactation stage, and pumping time. Differences are particularly observed between day and night breast milk in terms of circadian rhythms. Daytime milk contains higher levels of substances such as immune system-related nucleotides, interleukins, and antioxidants, while nighttime milk is rich in sleep-regulating components such as melatonin and tryptophan. This difference is important for the transmission of the mother's biological rhythms to the baby, contributing to the regulation of the baby's sleep-wake cycle and improving its environmental adaptation.

The chronobiological feeding model suggests that expressed breast milk be given in periods of day and night, or more specifically, in six-hour cycles, in accordance with the daily cycle. This approach aims to support the development of the infant's circadian rhythm through expressed breast milk in situations where breastfeeding is not possible. A review of the literature revealed no studies that combined PIOMI with chronobiological feeding. Therefore, this research was planned to determine the effects of oral motor intervention (PIOMI) and chronobiological feeding on feeding readiness, transition to total oral feeding and body weight in preterm infants hospitalized in the NICU.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants with a postnatal age of 29-33 weeks,
* Whose vital signs and clinical condition have been stable for at least 24 hours,
* Whose APGAR score at 1 and 5 minutes (Activity-Pulse-Grimace-Appearance-Respiration) is 4 or higher.

Exclusion Criteria:

* Infants with major congenital anomalies (such as congenital heart disease, cleft palate, cleft lip) or birth trauma,
* Infants with RDS,
* Infants diagnosed with asphyxia,
* Infants with intraventricular hemorrhage,
* Infants with Neonatal Withdrawal Syndrome,
* Infants with Fetal Alcohol Syndrome,
* Infants included in the study group who develop any complications or whose stable condition deteriorates during the follow-up period,
* Infants with feeding intolerance or who are interrupted from feeding for more than 48 hours,
* Infants who develop sepsis,
* Infants who develop necrotizing enterocolitis,
* Infants receiving mechanical ventilation support,
* Infants who receive narcotic analgesia or sedation,

Ages: 29 Weeks to 33 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 54 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Readiness for Feeding | Newborns At 29-33 Gestatıonal Weeks
  On days 1, 8, 11, and 14 of the study, the readiness of the infants for oral feeding will be assessed using the Premature Infant Readiness for Oral Feeding Assessment Scale. The Turkish validity and reliability of this scale, developed by Çamur and Çetinkaya, shows a cutoff point of 29. The maximum possible score on the scale is 36. A higher score indicates better readiness.
Transitioning to Total Oral Feeding | Newborns at 29-33 Gestatıonal Weeks
  Infants' nutritional information will be assessed daily using an infant monitoring form.
Body Weight | Newborns at 29-33 Gestatıonal Weeks
  Infants' body weights will be measured on days 1, 8, 11, and 14, on the day they start total oral feeding, and on the day they are discharged, at 8:30 AM, wearing only a clean diaper.

CONTACTS AND LOCATIONS:
Locations (1):
- Aydın Adnan Menderes University, Faculty of Nursing, Department of Child Health and Disease Nursing, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request
Supporting Information: Study Protocol
Time Frame: 6 months after publication
Access Criteria: relevance to the topic of the study and approval of all co-authors within 1 month of receiving the request.